CLINICAL TRIAL: NCT04195373
Title: A Phase I Open-label, Safety Study of Intra-tumoral Application of TMV-018 in Combination With 5-FC or Anti-PD-1 Therapy in Patients With Tumors of the Gastrointestinal Tract
Brief Title: A Safety Study of TMV-018 in Patients With Tumors of the Gastrointestinal Tract
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study not started, no subjects recruited.
Sponsor: Themis Bioscience GmbH (Industry)
Collaborators: Assign Data Management and Biostatistics GmbH (Other); Optimapharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMV-018-101
Record Dates: First submitted 2019-12-05; First posted 2019-12-11 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Gastrointestinal Cancer
Keywords: Colorectal cancer; Esophageal cancer; Gastric cancer; TMV-018; anti-PD-1; 5-FC; oncolytic virus
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMV-018 + 5-FC (Experimental): Patients will receive intra-tumoral TMV-018 on days 0, 14, 28 and 42, and will be additionally treated with the prodrug 5-FC.
  Interventions: Biological: TMV-018 + 5-FC
- TMV-018 + anti-PD-1 inhibitor (Experimental): Patients will receive intra-tumoral TMV-018 on days 0, 14, 28 and 42, and will be additionally treated with an anti-PD-1 Inhibitor.
  Interventions: Biological: TMV-018 + anti-PD-1
- TMV-018 + 5-FC + anti-PD-1 inhibitor (Experimental): Patients will receive intra-tumoral TMV-018 on days 0, 14, 28 and 42, and will be additionally treated with the prodrug 5-FC and an anti-PD-1 Inhibitor.
  Interventions: Biological: TMV-018 + 5-FC + anti-PD-1

INTERVENTIONS:
Biological: TMV-018 + 5-FC — TMV-018: liquid frozen, life attenuated, oncolytic measles virus encoding the prodrug converting enzyme "super cytosine deaminase"; 1E+06 TCID50 to 1E+08 TCID50 per dose.
  5-FC: 150 mg/kg/day for 2 days during each treatment.
  Arms: TMV-018 + 5-FC
Biological: TMV-018 + anti-PD-1 — TMV-018: liquid frozen, life attenuated, oncolytic measles virus encoding the prodrug converting enzyme "super cytosine deaminase"; 1E+06 TCID50 to 1E+08 TCID50 per dose.
  Anti-PD-1 inhibitor dose according to its SMPC.
  Arms: TMV-018 + anti-PD-1 inhibitor
Biological: TMV-018 + 5-FC + anti-PD-1 — TMV-018: liquid frozen, life attenuated, oncolytic measles virus encoding the prodrug converting enzyme "super cytosine deaminase"; 1E+06 TCID50 to 1E+08 TCID50 per dose.
  5-FC: 150 mg/kg/day for 2 days during each treatment cycle.
  Anti-PD-1 Inhibitor: dose according to its SMPC.
  Arms: TMV-018 + 5-FC + anti-PD-1 inhibitor

SUMMARY:
This study aims to determine the safety and tolerability of TMV-018 when given alone or in combination with the prodrug 5-Fluorocytosine (5-FC) or an anti-PD-1 checkpoint inhibitor in patients with gastrointestinal tumors. Furthermore, the maximum tolerated dose (MTD) and recommended Phase II dose of TMV-018 shall be determined.

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalation phase I trial that aims to determine the safety and tolerability of TMV-018, an oncolytic measles virus encoding the prodrug converting enzyme "super cytosine deaminase", when given alone or in combination with the prodrug 5-Fluorocytosine (5-FC) or an anti-PD-1 checkpoint inhibitor up to day 72 in patients with colorectal carcinoma (left-sided or rectal), esophageal carcinoma, or gastric cancer. Furthermore, the maximum tolerated dose (MTD) and recommended Phase II dose of TMV-018 shall be determined.

At least 15 patients will be enrolled. Patients will be randomized to different treatment groups: all patients will receive intra-tumoral TMV-018 on four visits and additionally 5-FC and/or anti-PD-1 treatment. All adverse events will be documented and analyzed for the primary safety endpoint. Blood and tumor samples will be collected up to day 72 to determine the safety, tolerability and immunogenicity of the treatment. The patients will be followed-up for another two years to determine long-term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any research procedures.
2. At least 18 years of age on the day of signing the informed consent.
3. Histologically confirmed diagnosis of advanced, metastatic tumors of the gastrointestinal tract (stage IV)
4. Before enrollment (i.e., at least 4 weeks before study treatment): Prior chemotherapy, targeted therapy, radiotherapy, to treat cancer or major surgery have to be stopped at least 4 weeks prior to enrolment.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and life expectancy ≥ 3 months as assessed during screening period.
6. All female participants of childbearing potential, defined as all woman physiologically capable of becoming pregnant, must have a negative pregnancy test at screening.
7. Willingness not to become pregnant or to father a child during study participation by practicing reliable methods of contraception.
8. Patient must have exhausted all current standard therapy lines in the target cancer indications
9. Adequate organ function as determined by laboratory parameters.

Exclusion Criteria:

1. Patients who participated in other studies of anti-tumor therapy within 2 weeks before enrolment.
2. Patients with brain metastases.
3. Patients with poorly controlled hypertension, or cardiovascular and cerebrovascular diseases with clinical significance.
4. Patients with other serious organic diseases or mental disorders.
5. Patients with active infections, which cannot be controlled with drugs or have potential impact on treatment, or patients with concurrent opportunistic infections.
6. Patients exhibiting evidence of clinically significant immunosuppression such as primary or acquired immunodeficiency state
7. Pregnancy (positive pregnancy test at screening or before end of study participation) or lactation at screening or planning to become pregnant before completion of study participation.
8. Males who have sex to conceive a child / who want to donate semen, during the study and up to 4 months after the last dose of TMV-018, 5-FC or pembrolizumab.
9. Males and female subjects of childbearing potential who are unwilling to use double barrier methods of effective contraception
10. Patients with an impaired renal function (creatinine clearance ≤ 40 mL/min).
11. Patients currently or recently (< 2 months) taking fluconazole, itraconazole, clotrimazole troches, itraconazole, amphotericin or other oral anti-fungal medications.
12. Patients with contraindications for treatment with flucytosine (5-FC)
13. Known hypersensitivity to 5-FU, known deficiency in dihydropyrimidine dehydrogenase (DPD)
14. Known hypersensitivity to pembrolizumab, its excipients, or other monoclonal antibody.
15. Severe immune-related adverse reactions from treatment with pembrolizumab, defined as any grade 4 toxicity or grade 3 toxicity requiring corticosteroid treatment (> 10 mg/day prednisone or equivalent) for greater than 12 weeks.
16. History or evidence of symptomatic autoimmune diseases.
17. Other medical condition or laboratory abnormality that in the judgment of the Investigator may increase the risk associated with study participation or may interfere with interpretation of study results.
18. History of severe systemic reaction or side-effect after a measles vaccination.
19. Subjects who continue to experience > grade 1 Common Terminology Criteria for Adverse Events (CTCAE) toxicity due to cancer therapy within 4 weeks prior to enrollment will not be eligible.
20. Use of anti-cancer treatments within 4 weeks of TMV-018 treatment start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 4 years
  Incidence of solicited and unsolicited adverse events from enrollment until end of study.
Determine MTD and dose for phase II | 1.5 years
  Determine the maximum tolerated dose (MTD) and recommended Phase II dose of TMV-018

SECONDARY OUTCOMES:
Viral replication | 2 years
  Assess viral replication at injected tumor sites, viremia (distribution of i.t. applied TMV-018 into the blood stream), and shedding as well as possible persistence phenomena of TMV-018
Viral distribution | 2 years
  Assess viremia (distribution of i.t. applied TMV-018 into the blood stream) and shedding as well as possible persistence phenomena of TMV-018
Efficacy of therapy assessed by RECIST 1.1 | 4 years
  Assess the therapeutic efficacy of TMV-018 with 5-FC or anti-PD-1 therapy by radiologic assessment (RECIST 1.1, time to progression).
Efficacy of therapy assessed by changes in tumor marker level | 4 years
  Assess the therapeutic efficacy of TMV-018 with 5-FC or anti-PD-1 therapy by changes in tumor marker level.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Lauer, MD, Principal Investigator — University Hospital Tuebingen
Locations (2):
- Germany (2):
  - University Hospital Bonn, Bonn
  - University Hospital Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No